CLINICAL TRIAL: NCT04773301
Title: Randomized and Controlled Phase IV Clinical Trial on the Analgesic Effectiveness of the Combined Blockade in the Hip Fractures of the Elderly: Comparative Study Between Levobupivacaine and Ropivacaine
Brief Title: Comparative Study Between Levobupivacaine and Ropivacaine in the Hip Fractures of the Elderly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León (Other)
Collaborators: Instituto de Investigación Biomédica de Salamanca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PENG-CAD; 2020-004697-21 (EudraCT Number)
Record Dates: First submitted 2021-02-15; First posted 2021-02-26 (Actual); Results first posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Levobupivacaine; Ropivacaine

STUDY DESIGN:
Intervention Model Description: Low-intervention clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LEVOBUPIVACAINE (Experimental): Patients treated with Levobupivacaine Altan 7.5 mg / ml solution for injection and infusion
  Interventions: Drug: Levobupivacaine
- ROPIVACAINE (Experimental): Patients treated with Ropivacaine Altan 2 mg / ml solution for infusion
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Levobupivacaine — Local anaesthetic drug belonging to the amino amide group. It is the S-enantiomer of bupivacaine
  Other Names: Levobupivacaína Altan 7,5 mg/ml solución inyectable y para perfusión E F G
  Arms: LEVOBUPIVACAINE
Drug: Ropivacaine — Local anaesthetic drug belonging to the amino amide group. The name ropivacaine refers to both the racemate and the marketed S-enantiomer.
  Other Names: Ropivacaína Altan 2 mg/ml solución para perfusión EFG
  Arms: ROPIVACAINE

SUMMARY:
Prospective, low-level, non-commercial intervention, comparative clinical trial (phase IV) of balanced, randomized groups, to compare the analgesic efficacy of the local anesthetics Ropivacaine and Levobupivacaine in peripheral nerve block in hip fracture surgery in the elderly .

DETAILED DESCRIPTION:
There are several studies that try to identify the ideal anesthetic for the management and control of pain in hip fracture surgery in the elderly. The optimum would be to use an anesthetic with the lowest possible latency, since this will favor the start of surgery. And, at the same time, with a more lasting analgesia with the least motor impairment. Therefore, it is essential to collect data on efficacy (effective block that allows us to mobilize the patient), latency, and analgesic scales appropriate to the cognitive state of the study sample.

ELIGIBILITY:
Inclusion Criteria:

* The patient will have to voluntarily sign and understand the informed consent that will be provided in writing.
* Patients over 65 years of age, with a hip fracture, who are going to be operated on at the Salamanca University Assistance Complex (CAUSA).

Exclusion Criteria:

* Rejection of the technique.
* Allergy to any of the drugs.
* Coagulation disorders.
* Local infections instead of puncture.
* Vascular prostheses at the femoral level.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 114 (Actual)
Dates: Start 2021-02-13 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Agustín Díaz Álvarez, MD PhD, Principal Investigator — University of Salamanca
Locations (1):
- Complejo Asistencial Universitario de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Salgado-Garcia D, Diaz-Alvarez A, Gonzalez-Rodriguez JL, Lopez-Iglesias MR, Sanchez-Lopez E, Sanchez-Ledesma MJ, Martinez-Trufero MI. Comparison of the Analgesic Efficacy between Levobupivacaine 0.25% and Ropivacaine 0.375% for PENG (Pericapsular Nerve Group) Block in the Context of Hip Fracture Surgery of Elderly Patients: A Single-Center, Randomized, and Controlled Clinical Trial. J Clin Med. 2024 Jan 29;13(3):770. doi: 10.3390/jcm13030770. PMID 38337464

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LEVOBUPIVACAINE | ROPIVACAINE
Started | 57 | 57
Completed | 56 | 52
Not Completed | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LEVOBUPIVACAINE | ROPIVACAINE | Total
Number analyzed (Participants) | 56 | 52 | 108
Age, Continuous [Median (Standard Deviation); unit: years] | 86.40 (7.56) | 86.13 (8.47) | 86.27 (7.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 43 | 84
  Male | 15 | 9 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Spain | 56 | 52 | 108
Patients Treated [Count of Participants; unit: Participants] | 56 | 52 | 108

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of the Analgesic Efficacy of Both Local Anesthetics in the Regional Block of Hip Fracture Surgery
Description: The primary measure of efficacy in this study will be the difference in block duration. To evaluate this, the need for rescue medication will be assessed at several time points, including 6, 12, 24, and 48 hours.
Time Frame: 6h, 12h, 24h and 48h
Measure: Count of Participants; unit: Participants
Arm/Group | LEVOBUPIVACAINE | ROPIVACAINE
Number analyzed (Participants) | 56 | 52
Participants
  6h | 10 | 4
  12h | 12 | 14
  24h | 21 | 17
  48h | 10 | 14
  No rescue | 3 | 3

2. Secondary Outcome: Latency of Initiation.
Description: This study aims to describe the behavior of the combined technique in hip fractures by establishing the latency of initiation.
  Latency: evaluated by analgesic scales up to 48 hours. Analgesic scales: EVN - numerical verbal scale- (0= No pain (min) - 10=The worst pain imaginable (max)), Algoplus (0=min - 5=max) and PAINAD -Paint Assessment in Advanced Dementia- (0=min - 10=Max). They will be carried out at 6, 12, 24 and 48 h after the procedure blocking. In both scales, the lowest values are those of better outcome and the highest are those of worst outcome.
  Need and rescue drugs: rescue analgesia will be prescribed for the hospital ward, in case it is necessary. The need, drug and time of administration will be collected regarding the execution of the blockade.
Time Frame: The duration of treatment for each patient will be considered until the evaluation of the analgesic scale corresponding to 48 hours after the procedure is performed.
Population: EVN, ALGOPLUS and PAINAD pain rating scales in patients treated with Levobupivacaine or Ropivacaine
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- EVN Scale - LEVOBUPIVACAINE: Patients treated with Levobupivacaine Altan 7.5 mg / ml solution for injection and infusion
  Levobupivacaine: Local anaesthetic drug belonging to the amino amide group. It is the S-enantiomer of bupivacaine
  Numerical Visual Scale (EVN): (0= No pain (min) - 10=The worst pain imaginable (max))
- EVN - Scale ROPIVACAINE: Patients treated with Ropivacaine Altan 2 mg / ml solution for infusion
  Ropivacaine: Local anaesthetic drug belonging to the amino amide group. The name ropivacaine refers to both the racemate and the marketed S-enantiomer.
  Numerical Visual Scale (EVN): (0= No pain (min) - 10=The worst pain imaginable (max))
- ALGOPLUS Scale - LEVOBUPIVACAINE: Patients treated with Levobupivacaine Altan 7.5 mg / ml solution for injection and infusion
  Levobupivacaine: Local anaesthetic drug belonging to the amino amide group. It is the S-enantiomer of bupivacaine
  Algoplus Scale (ALGSC): Face, looks, complaints, body and behavior. 0=Min - 5=Max
- ALGOPLUS Scale - ROPIVACAINE: Patients treated with Ropivacaine Altan 2 mg / ml solution for infusion
  Ropivacaine: Local anaesthetic drug belonging to the amino amide group. The name ropivacaine refers to both the racemate and the marketed S-enantiomer.
  Algoplus Scale (ALGSC): Face, looks, complaints, body and behavior. 0=Min - 5=Max
- PAINAD Scale - LEVOBUPIVACAINE: Patients treated with Levobupivacaine Altan 7.5 mg / ml solution for injection and infusion
  Levobupivacaine: Local anaesthetic drug belonging to the amino amide group. It is the S-enantiomer of bupivacaine
  Paint Assessment in Advanced Dementia Scale (PAINAD):Breathing (independent of vocalization), Negative vocalization, Facial expression, Body language and Consolability. 0=Min - 10=Max
- PAINAD Scale - ROPIVACAINE: Patients treated with Ropivacaine Altan 2 mg / ml solution for infusion
  Ropivacaine: Local anaesthetic drug belonging to the amino amide group. The name ropivacaine refers to both the racemate and the marketed S-enantiomer.
  Paint Assessment in Advanced Dementia Scale (PAINAD):Breathing (independent of vocalization), Negative vocalization, Facial expression, Body language and Consolability. 0=Min - 10=Max
Arm/Group | EVN Scale - LEVOBUPIVACAINE | EVN - Scale ROPIVACAINE | ALGOPLUS Scale - LEVOBUPIVACAINE | ALGOPLUS Scale - ROPIVACAINE | PAINAD Scale - LEVOBUPIVACAINE | PAINAD Scale - ROPIVACAINE
Number analyzed (Participants) | 56 | 52 | 56 | 52 | 56 | 52
score on a scale
  6h | 1.92 (1.04) | 1.68 (2.56) | 0.94 (1.25) | 0.75 (1.04) | 1.46 (2.05) | 1.04 (1.67)
  12h | 2.50 (2.26) | 2.91 (3.15) | 1.3 (1.06) | 1.38 (1.43) | 1.95 (1.69) | 1.84 (1.99)
  24h | 4.33 (2.79) | 3.5 (2.82) | 2.16 (1.37) | 1.70 (1.28) | 3.22 (1.99) | 2.76 (2.17)
  48h | 4.72 (2.66) | 4.58 (2.84) | 2.32 (1.27) | 2.21 (1.33) | 3.75 (2.33) | 3.36 (2.14)

3. Secondary Outcome: Secondary Effects Derived From the Combined Technique Described.
Description: Number of participants with treatment-related adverse events as assessed by CTCAE version 5.0 will be used to report toxicity and adverse events.
Time Frame: as for outcome 2
Reporting Status: Not Posted

4. Secondary Outcome: Usefulness of the Chosen Analgesic Scale in Our Population, Especially in Patients With Cognitive Impairment.
Description: We will use 3 assessment scales:
  Numerical Visual Scale (EVN): 0=No pain - 5=The worst pain imaginable Algoplus Scale (ALGSC): Face, looks, complaints, body and behavior. 0=Min - 5=Max Paint Assessment in Advanced Dementia Scale (PAINAD):Breathing (independent of vocalization), Negative vocalization, Facial expression, Body language and Consolability. 0=Min - 5=Max
Time Frame: as for outcome 2
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: At 48 h it is considered the end of follow-up
Arm/Group | LEVOBUPIVACAINE | ROPIVACAINE
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/52
Other Adverse Events (participants affected / at risk) | 0/56 | 0/52

LIMITATIONS AND CAVEATS:
The age of the patients often makes it difficult for researchers to interpret pain scales.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT04773301/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT04773301/ICF_001.pdf